CLINICAL TRIAL: NCT01825733
Title: Comparison of Palonosetron and Ramosetron for Preventing Patient-controlled Analgesia Related Nausea and Vomiting Following Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2011-0122
Record Dates: First submitted 2013-03-26; First posted 2013-04-08 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: palonosetron, ramosetron, PONV, opioid
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ramosetron; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ramosetron (Experimental)
  Interventions: Drug: ramosetron
- palonosetron (Active Comparator)
  Interventions: Drug: palonosetron

INTERVENTIONS:
Drug: ramosetron — Ramosetron 0.3 mg was mixed to the PCA. Same dose of drug was administered 10 minutes before the end of surgery according to the allocated group.
  Arms: ramosetron
Drug: palonosetron — palonosetrno 0.075 mg was mixed to the PCA. Same dose of drug was administered 10 minutes before the end of surgery according to the allocated group.
  Arms: palonosetron

SUMMARY:
Postoperative pain, the great concern for the patients undergoing spine surgery, has led to common use of opioid-based intravenous patient-controlled analgesia (IV-PCA) postoperatively. Opioid-based IV-PCA offers better pain control, which could facilitate early recovery, rehabilitation and increase patient satisfaction. However, its use inevitably increases the incidence of postoperative nausea and vomiting (PONV), another great discomfort, as high as 80% in patients with multiple risk factors.Therefore, there have been consistent efforts to prevent PONV with multimodal therapies such as risk stratification, modification and preventive use of antiemetics.

Of all antiemetics, 5-hydroxytryptamine (5-HT3) antagonist, especially ondansetron, is most commonly used and extensively studied to reduce PONV because of its efficacy and fewer side effects.[8] However, its efficacy is not quite satisfactory when it comes to PONV associated with opioid-based IV-PCA. Recently, there are many reports comparing the antiemetic efficacy between ondansetron and the 2 newly developed 5-HT3 antagonists, ramosetron and palonosetron. Ramosetron is known to have a higher affinity and longer duration of binding to 5-HT3 receptor, therefore exhibits potent and sustained anti-emetic effect than previously developed 5-HT3 antagonists.Palonosetron has a unique allosteric binding to the 5-HT3 receptor, which brings a higher affinity, longer duration of action and longer elimination half-time.According to the previous studies, both ramosetron and palonosetron showed superior antiemetic efficacy for PONV associated with opioid-based IV-PCA to ondansetron as expected by their theoretical advantages. However, it has never been evaluated which one has superior antiemetic efficacy for opioid-based IV-PCA associated PONV. Therefore, in this study, we tried to evaluate the relative antiemetic efficacy of ramosetron and palonosetron in controlling opioid-based IV-PCA related PONV.

ELIGIBILITY:
Inclusion Criteria:

1. patients (20-65 years) scheduled for lumbar spinal surgery in prone position between August 2011 and July 2012.
2. All patients were using opioid-based IV-PCA postoperatively for pain control

Exclusion Criteria:

1. gastrointestinal disease
2. renal dysfunction
3. hepatic dysfunction
4. diabetes mellitus on insulin
5. pregnancy
6. use of steroid, opioid, antiemetics within 1 day before surgery
7. inability to understand verbal rating scale (VRS)
8. inability to use PCA device

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
verbal numeric scale | change of antiemetic efficacy for 5 time points ( postanesthesia care unit, 0-6 h, 6-24 h, 24-48 h, 48-72 h after operation)
  At each time point, frequency and intensity (verbal numeric scale, 0-10, 0: no nausea, 10: maximum) of nausea, frequency of vomiting, rescue antiemetic use were recorded and compared between groups.